CLINICAL TRIAL: NCT05445141
Title: Little ACF: A Randomized Controlled Trial on Effects of Universal Parental Group Support Regarding Infants Aged 12-24 Months
Brief Title: Little ACF (Lilla ABC): Evaluation of a Parental Support Program for Parents of Children Aged 1-2 Years
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Lene Lindberg, Associate Professor in Psychology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VR Dnr: 2021-06447
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Parental Support; Emotion Regulation; Coping Behavior; Stress, Emotional; Coparenting
MeSH Terms: conditions — Emotional Regulation; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The study is a two-armed study including an intervention group and a control group. The groups consist of parents of children 1-2 years that are registered at any of the included CHCs in the study.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Parents included in the intervention group will be offered to participate in four meetings that are taking place during four weeks time. The focus of the meetings is on how to promote parent-infant relationship. The theoretical base is positive developmental psychology including research on attachment, parenting and co-parenting, emotional regulation, and observational learning/role models. Roleplays, video-clips, discussions, and individual reflections are used to empower families during the sessions. Parents are encouraged to try the content with their child between the sessions and will be provided a printed material.
  Interventions: Behavioral: Little ACF [in Swedish: Lilla ABC]
- Control (Sham Comparator): Parents in the control group will via a web-based portal be able to view four pre-recorded lectures during four weeks. The lectures will be around 10 minutes long and have a content similar to the group meetings that are offered to the intervention group but more superficial and without printed material and reflection practices.
  Interventions: Behavioral: Lectures

INTERVENTIONS:
Behavioral: Little ACF [in Swedish: Lilla ABC] — Little ACF is a modified version of the program called All Children in Focus [in Swedish: Alla Barn i Centrum (ABC)] that originally is developed for parents with children 3-12 years of age. The content is based on positive developmental psychology and involves role plays, discussions and exercises to try at home with the child. Printed material will be provided to the parents at each meeting/session. Little ACF is offered once a week during four weeks. Each session is 60 minutes, thereafter the parents can stay in the facility for 30 minutes to continue discussing with each other.
  Arms: Intervention
Behavioral: Lectures — The lectures are pre-recorded and available during four weeks. Each lecture is 10 minutes and the content is similar to, but more superficial than, the content in Little ACF.
  Arms: Control

SUMMARY:
Society can promote children's mental health at an early stage by creating good conditions with, for example, general parental support programs that are offered to all parents. One program that has been developed is called All Children in Focus (ACF) [in Swedish: Alla Barn i Centrum (ABC)] which has been evaluated for parents with children aged 3-12 years. The results showed effects on parenting ability, parenting strategies and on children's well-being. Staff in child health care (CHC), a natural arena for parental support programs reaching almost all families, have requested modifications in the program ACF to involve parents with younger children. The parent groups offered within CHC today are not evaluated in younger children and could be thus replaced by researched parental support based on evidence.

The investigators therefore want to study the effects of a modified version of ACF for parents of children 1-2 years (Little ACF) to see if Little ACF can strengthen parenting ability and have effects on children's social and emotional development. Parents within CHC are asked to participate and are randomly assigned to Little ACF or the regular CHC program plus a lecture. Little ACF is offered during four group meetings and potential effects are measured with questionnaires. Measurements are made before randomisation, during and after participation in Little ACF. Children's behavior is followed up at 3 years through questionnaires and CHC documentation.

The study can provide important knowledge about how Little ACF can promote children's mental health and strengthen parents. The investigators see it as a strength that Little ACF is based on research and on dialogue with parents and professionals. Little ACF, which is aimed at everyone, can form a basis for identifying families and children who need preventive and treatment measures.

DETAILED DESCRIPTION:
Promotion of mental health is an important topic and early interventions may be the most cost-effective investment for the society. The Child Health Care (CHC) in Sweden reaches 99% of parents with infants and is the society's major promotive support during the first years of life. All Children in Focus (ACF) [in Swedish: Alla Barn i Centrum (ABC)] is a universal program aiming to support positive parental strategies and promote child well-being. ACF has shown positive effects for parental efficacy and strategies and for child well-being at age 3-12 years. In this 3-year project the investigators aim to gain knowledge about how ACF given to parents with children 1-2 years (Little ACF) may influence parenting and child well-being. Specific research questions are how Little ACF in comparison to care as usual (CAU) within CHC can:

* strengthen strategies of emotional regulation in parents,
* promote parenting practices,
* promote child well-being
* lead to reduction of child behavior problems (externalizing/internalizing),
* engage and retain parents in groups?

Parents with infants of 12-24 months that are registered at any of the included CHC centers in Stockholm, Gotland and mid-Sweden will be asked for participation. Recruitment will be performed at the ordinary 10-, 12- or 18-months visits of the child. The CHC nurse will ask parent/s for participation verbally and parents will be provided the information and consent form and a pamphlet about the study. Parents who are interested in participating will be sent a link via email with the same information and consent form that can be signed digitally. Thereafter they will be sent the questionnaire. When the CHC nurse has recruited twice as many parents as a full Little ACF group, the researchers will randomize the parents into the two groups, one receiving the intervention Little ACF and the other a control group receiving CAU and digital lectures. The CHC nurse will notify the parents about which group they have been randomized to and a description on how the study will proceed.

A previous randomized study of ACF (aimed at parents with children 3-12 years) showed an effect size (Cohen's d) of 0.30 for parental self-efficacy. Since this study compares Little ACF with CAU including lectures (instead of waiting list), a marginally smaller effect (d = 0.25) between the groups is expected. With a significance level of 95% (p-value 0.05) and a power of 80%, it would thus be needed 251 participants in each group. A drop-out rate of 25% is expected, which means that a total of 670 families would need to be included.

Each Little ACF group will consist of parents of 5-7 children, which means that about 60-70 groups will be needed and thus a total of 25 group leader pairs if each pair leads three groups. The pair of group leaders consist of one CHC nurse and one social worker or other profession with experience of working with parents of young children. Group leaders will be provided a training containing theory, practical exercises, and supervision. The training is spread out over three occasions taking place every other week to allow for the possibility to start Little ACF groups in between the training sessions. After the training, the group leaders will be offered monthly group supervision.

Effects of Little ACF on positive parenting and strategies are assessed through parental questionnaires distributed digitally to be completed independently by the parents. Child well-being is measured through parental questionnaires and data in CHC records. CHC nurses will be invited to semi-structured interviews to gain a better knowledge in how the experience of Little ACF affect daily work at CHC. Quantitative data will be analyzed statistically with linear regression models and qualitative data will be analyzed using thematic analysis.

This study adds to the evidence of promotion during infancy and give information if Little ACF is effective for parents and young children. It may also reduce needs of future interventions of mental health problems.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children in the age of 1-2 years that are registered at the CHCs included in the study

Exclusion Criteria:

* Parents in need of interpreter will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in parental self-efficacy from baseline to four different time points: directly after the intervention, after 6 months, 12 months and when the child is 3 years old. | At five occations: baseline (T1), directly after the intervention (T2), after 6 months (T3), 12 months (T4) and in relation to the child's visit to CHC at 3 years of age (T5))
  Will be measured with the "Tool to Measure Parenting Self-Efficacy" - TOPSE (Bloomfield & Kendall, 2012), with 48 statements that are to be answered to on a 11 point scale, from 0=not agree to 10=fully agree
Change in parent emotion regulation from baseline to four different time points: directly after the intervention, after 6 months, 12 months and when the child is 3 years old. | At five occations: baseline (T1), directly after the intervention (T2), after 6 months (T3), 12 months (T4) and in relation to the child's visit to CHC at 3 years of age (T5))
  Will be measured with the "Parent Emotion Regulation Scale" - PERS (Pereira et al., 2017). The scale has 20 statements that should be rated on a 5-point scale, from 1=never or almost never to 5=always or almost always.
Change in coping with the negative emotions of the child from baseline to four different time points: directly after the intervention, after 6 months, 12 months and when the child is 3 years old. | At five occations: baseline (T1), directly after the intervention (T2), after 6 months (T3), 12 months (T4) and in relation to the child's visit to CHC at 3 years of age (T5))
  Will be measured using "Coping with Toddlers' Negative Emotion Scale" - CTNES (Spinrad et al, 2007), the scale has 12 scenarios with 7 options each on how a parent would react that to that specific scenario (Distress reactions, Punitive reactions, Expressive encouragement, Emotion-focused reactions, Problem-focused reactions, Minimization reactions and Granting wish reactions), the parent are asked to rate how likely s/he is to react in that specific manner from 1 = very unlikely to 7 = very likely, the higher the score the more likely to use that coping mechanism.
Change in parental stress from baseline to four different time points: directly after the intervention, after 6 months, 12 months and when the child is 3 years old. | At five occations: baseline (T1), directly after the intervention (T2), after 6 months (T3), 12 months (T4) and in relation to the child's visit to CHC at 3 years of age (T5))
  Will be measured using the scales (1) incompetence, (2) social isolation and (3) role restriction from the "Swedish Parenting Stress Questionnaire" - SPSQ (Östberg, Hagekull & Wettergren, 1997), the scale is from 1 to 5 indicating 'Strongly disagree' to 'Strongly agree', the total possible score is 170 and higher scores indicate higher stress.
Change in coparenting relationship from baseline to four different time points: directly after the intervention, after 6 months, 12 months and when the child is 3 years old. | At five occations: baseline (T1), directly after the intervention (T2), after 6 months (T3), 12 months (T4) and in relation to the child's visit to CHC at 3 years of age (T5))
  Will be measured using 5 items from "The Coparenting Relationship Scale" (Feinberg et al., 2012), to be answered with a 5 point scale from 1=not agree to 5=fully agree

SECONDARY OUTCOMES:
Change in childrens' social and emotional development from baseline to four different time points: directly after the intervention, after 6 months, 12 months and when the child is 3 years old. | At five occations: baseline (T1), directly after the intervention (T2), after 6 months (T3), 12 months (T4) and in relation to the child's visit to CHC at 3 years of age (T5), expected effect at T3, T4 and T5
  Will be measured using "Ages & Stages Questionnaires - Socio-Emotional Second Edition" (ASQ: SE-2; Singh et al., 2017)
Psychological and behavioural problems | In relation to the child's visit to CHC at 3 years of age (T5), expected effect at T5
  Strength and Difficulties Questionnaire (SDQ; Theunissen et al., 2013) that is being sent out before the child's visit to CHC at 3 years of age and that is registered in CSAM Health Analytics (medical record system at CHC).

CONTACTS AND LOCATIONS:
Overall Officials: Lene Lindberg, Ass Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Central Child Health Care (Centrala barnhälsovården), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blom L, Edenius A, Enebrink P, Hjern A, Silfverdal SA, Ahlen J, Bergstrom M, Lindberg L. Little All Children in Focus (Little ACF), evaluation of a parental support program for parents of children aged 1-2 years: study protocol for a randomized controlled trial. Trials. 2023 Mar 13;24(1):184. doi: 10.1186/s13063-023-07212-4. PMID 36907876